CLINICAL TRIAL: NCT06424600
Title: Effect of Various Forms of Nicotine Consumption on Gingival Health of Dental Patients.
Brief Title: Ginglival Health Among Smokers Visiting Dental Hospital
Status: Completed | Type: Observational
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Afsheen Mansoor, Principle Investigator, Pakistan Institute of Medical Sciences
Other Study IDs: SOD/ERB/2023/32-02
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Smoking
Keywords: Gingival; Smokers
MeSH Terms: conditions — Smoking | interventions — Periodontal Index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- S-form users: Smoke- form users
  Interventions: Other: Gingival Index
- E-form users: E-Cigarette users
  Interventions: Other: Gingival Index
- D-form users: Dual-Form users
  Interventions: Other: Gingival Index

INTERVENTIONS:
Other: Gingival Index — The G-I index ranging between 0.5-2 was used to calculate the occurrence of severe gingival issues in participants with smoking habits. The G-I index between 0.50-1.00 displayed light gingival inflammation, G-I between 1.10-2.00 revealed moderate gingival inflammation and G-I > 2.00 confirmed severe gingival inflammation.

SUMMARY:
The effect of different forms of nicotine intake on the gingival health of dental patients that visited a public sector in Islamabad. A total of 300 dental patients that visited School of Dentistry, Islamabad voluntarily participated in this study. The nicotine consuming participants involved in this study were Smoke-form users, E cigarette-form users, and Dual-form users whose Gingival Index (G-I) was inspected to demonstrate an association between their smoking type and duration of developing severe gingivitis.

DETAILED DESCRIPTION:
A total of 300 dental patients who visited the School of Dentistry, Islamabad, participated voluntarily in this study. The nicotine-consuming participants involved in this study were Smoke-Form users (S-form), Electronic cigarette-form users (E-form), and Dual-Form users (D-form) whose Gingival Index (G-I) was inspected to demonstrate an association between their smoking type and duration of developing severe gingivitis. The G-I ranging between 0.5 - 2.00 was used to calculate the occurrence of severe gingival issues in participants with smoking habits where G-I between 0.50 1.00 displayed Light gingival inflammation, G-I between 1.10-2.00 revealed Moderate gingival inflammation and G-I > 2.00 confirmed Severe gingival inflammation. A chi-Square test was used for the association by keeping significance p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Smokers with good general health status visiting dental hospital

Exclusion Criteria:

* Non-smoker dental patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting Dental Outpatient Department with history of Smoking
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Gingival Index | one year
  The G-I ranging between 0.5-2 was used to calculate the occurrence of severe gingival issues in participants with smoking habits where G-I between 0.50-1.00 displayed Light gingival inflammation, G-I between 1.10-2.00 revealed Moderate gingival inflammation and G-I > 2.00 confirmed Severe gingival inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Afsheen Mansoor, Principal Investigator — Pakistan Institute of Medical Sciences
Locations (1):
- Afsheen Mansoor, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomar SL, Hecht SS, Jaspers I, Gregory RL, Stepanov I. Oral Health Effects of Combusted and Smokeless Tobacco Products. Adv Dent Res. 2019 Oct;30(1):4-10. doi: 10.1177/0022034519872480. PMID 31538806